CLINICAL TRIAL: NCT03220269
Title: RIAC - Registro Italiano Arresti Cardiaci. An Observational, Prospective, Multi-centre, Study of Epidemiology, Treatment, and Outcome of Cardiac Arrest
Brief Title: RIAC - Registro Italiano Arresti Cardiaci (Italian Registry of Cardiac Arrest)
Acronym: RIAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Italian Resuscitation Council (Other)
Responsible Party: Sponsor
Other Study IDs: RIAC
Record Dates: First submitted 2017-06-22; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Out-Of-Hospital Cardiac Arrest; In-hospital Cardiac Arrest
Keywords: Utstein; Resuscitation; Epidemiology; Emergency medicine; Resuscitation Registry
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Out-of-hospital cardiac arrest (OHCA): An OHCA is defined as cessation of cardiac mechanical activity that occurs outside of the hospital setting and is confirmed by the absence of signs of circulation.
  Interventions: Other: Out-of-hospital cardiac arrest (OHCA)
- In-hospital cardiac arrest (IHCA): An IHCA is defined as cessation of cardiac mechanical activity that occurs inside of the hospital setting and is confirmed by the absence of signs of circulation.
  Interventions: Other: In-hospital cardiac arrest (IHCA)

INTERVENTIONS:
Other: Out-of-hospital cardiac arrest (OHCA) — Data collection
  Groups: Out-of-hospital cardiac arrest (OHCA)
Other: In-hospital cardiac arrest (IHCA) — Data collection
  Groups: In-hospital cardiac arrest (IHCA)

SUMMARY:
RIAC - An Observational, Prospective, Multi-centre, Study of Epidemiology, Treatment, and Outcome of Cardiac Arrest in Italy.

DETAILED DESCRIPTION:
The Italian Registry of Cardiac Arrest (RIAC) has been established in Italy by the Italian Resuscitation Council (IRC). It is a free web registry based on Utstein style data collection for all EMS and ICU departments that want to participate to this study.

This research project will include all events that occur between 00.00 on October 1st, 2014 and 23:59 on September 30th, 2019. The RIAC registry allows to follow and collect data from consecutive patients with cardiac arrest.

The expected outcomes of RIAC are:

* The implementation of an Italian registry of cardiac arrest that allows the prospective data collection.
* The study of the incidence of out-of-hospital cardiac arrest (OHCA) among the general population and related outcomes (hospital admission and long-term outcomes). An observational, prospective, multi-centre study on patients assisted by EMS which collect data on cardiac arrest using RIAC.
* The study of the incidence of in-hospital cardiac arrest (IHCA) among hospitalized patients, the quality level of treatments during the hospitalization period and the long-term outcomes. An observational, prospective, multi-centre study on hospitalized patients in hospitals which can efficaciously respond to an in-hospital emergency and collect data on cardiac arrest using RIAC.
* The study of the quality of post-resuscitation treatments for patients who suffered a cardiac arrest (OHCA-IHCA) admitted to ICUs. An observational, prospective, multi-centre study on patients admitted to ICUs which collect data on cardiac arrest using RIAC.
* A national database of cardiac arrest that will enable future participations to European projects, such as EuReCa "An international, prospective, multi-centre, three-month survey of epidemiology, treatment and outcome of patients suffering an out-of-hospital cardiac arrest in Europe".

For the perspective incidence study of IHCA, OHCA and the quality of post-resuscitation treatments, all cases with a cardiac arrest diagnosis aged ≥ 18 years old will be included. All patients without a cardiac arrest diagnosis will be excluded.

The main outcomes for the study population are listed for each subgroup.

Out-of-hospital Cardiac arrest:

* Estimate the incidence of cardiac arrest among the representative general population.
* Describe the implemented interventions outcomes.
* Define the cohort of out-of-hospital cardiac arrest arrived alive at the emergency department and describe the in-hospital pathway.
* Evaluate the quality of long-term outcomes (30-days survival; survival to discharge) of patients discharged alive.

In-hospital cardiac arrest:

• It is expected to enlist 10-20 patients per year per each participating hospital.

Quality of post-resuscitation treatments in ICUs:

• It is expected to enlist a number of patients which is calculated as the number of survived patients to IHCA and hospitalized in ICU plus the number of patients with OHCA arrived alive at emergency unit and hospitalized in ICU.

Statistical data analysis will be based on three main objectives. The incidence of cardiac arrest for OHCA will be evaluated as the ratio between the number of confirmed OHCA occurred during the whole study and the referring population.

The incidence of cardiac arrest for IHCA will be calculated using as denominator, the population at risk (ordinary recovery other than day hospital and day surgery). For the evaluation study of the quality level of treatments in Intensive Care Units, a multivariate analysis will be performed to assess the connection between outcomes and treatments. In particular, the relation between injury variable (duration of no-flow time and CPR defined as flow <20%), treatments (temperature, glycaemia, convulsions, hypothermia, serum potassium levels, acidosis during the first 72 hours, etc.) and outcome to discharge defined using CPC classification, will be evaluated.

The proportion of patients with CPC 3 and CPC 4 on the amount of IHCA an OHCA cardiac arrests, will be evaluated.

All participanting EMS/hospitals able to provide at least the core data, need to fill out a letter of intent to participate in this study and must provide an ethical approval from the local Ethical Committee.

ELIGIBILITY:
Inclusion Criteria:

All patients aged ≥ 18 years old who undergo an out-of-hospital cardiac or an in-hospital cardiac arrest.

Exclusion Criteria:

All patients without a cardiac arrest diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest patients
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence for OHCA and IHCA | Latest data inclusion December, 31st 2019
  The aim of the RIAC study is to determine the number of cardiac arrest for out-of hospital cardiac arrest and for in-hospital cardiac arrest events.
Outcome for OHCA and IHCA | Latest data inclusion March 31st, 2020
  The aim is to determine the percentage of Return of Spontaneous Circulation (ROSC) and six months survival with good neurological performance (assessed with Cerebral Performance Category scale) with a CPC score between 1-2, after 6 months of the cardiac arrest.

SECONDARY OUTCOMES:
30 days survival | Latest data inclusion December, 31st 2019
  Status of survival after 30 days after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Erga Cerchiari, MD, Principal Investigator — Department of Anesthesia and Intensive Care, Maggiore Hospital, AUSL, Bologna, Italy and Italian Resuscitation Council, Bologna, Italy; Giuseppe Ristagno, MD, PhD, Study Director — IRCCS-Istituto di Ricerche Farmacologiche "Mario Negri", Milan, Italy and Italian Resuscitation Council, Bologna, Italy; Federico Semeraro, MD, Study Director — Department of Anesthesia and Intensive Care, Maggiore Hospital, AUSL, Bologna, Italy and Italian Resuscitation Council, Bologna, Italy; Giovanni Gordini, MD, Principal Investigator — Department of Anesthesia and Intensive Care, Maggiore Hospital, AUSL, Bologna, Italy and Italian Resuscitation Council, Bologna, Italy
Locations (1):
- Italian Resuscitation Council, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for inclusion/participation in European cardiac arrest registries from European scientific societies or consortium, i.e. EuReCa registry from European Resuscitation Council. Data sets to be shared will be selected based on data required from the European registry. Data shared will be anonimized with no possibility to retrieve personal patient information. Data sharing will be approved by the RIAC Steering Committe and data will be transfered to the other Registry in a secure way under the direction of the Scientific Committee

REFERENCES:
- See also: RIAC official website — http://riac2014.ircouncil.it
- See also: IRC official website — http://www.ircouncil.it